CLINICAL TRIAL: NCT05452278
Title: A Randomised, Cross-over, Single-blind, Relative Bioavailability Study of Nicotine Delivery From Selected Oral Nicotine Products
Brief Title: A Relative Bioavailability Study of Nicotine Delivery From Selected Oral Nicotine Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial Brands PLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IB-OND-ZONEX-11
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Product sequence ABCD (Experimental): Subjects use Product A on Day 1, Product B on Day 2, Product C on Day 3 and Product D on Day 4
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D
- Product sequence BCDA (Experimental): Subjects use Product B on Day 1, Product C on Day 2, Product D on Day 3 and Product A on Day 4
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D
- Product sequence CDAB (Experimental): Subjects use Product C on Day 1, Product D on Day 2, Product A on Day 3 and Product B on Day 4
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D
- Product sequence DABC (Experimental): Subjects use Product D on Day 1, Product A on Day 2, Product B on Day 3 and Product C on Day 4
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D

INTERVENTIONS:
Other: Product A — Tobacco-free pouch, 14 mg nicotine/pouch, used for 20 minutes
Other: Product B — Tobacco-free pouch, 16 mg nicotine/pouch, used for 20 minutes
Other: Product C — Tobacco-free pouch, 20 mg nicotine/pouch, used for 20 minutes
Other: Product D — Tobacco pouch, 16.6 mg nicotine/pouch, used for 20 minutes

SUMMARY:
This will be a randomised, cross-over, single-blind, confinement study conducted in 27 male or female snus or nicotine pouch users. The study will investigate 4 different nicotine containing products in a cross-over design, incorporating pharmacokinetic (PK) evaluation, nicotine extraction evaluation, subjective questionnaire assessments as well as safety and tolerability evaluation.

During the study participation, subjects will come for 2 visits to the clinic, including a screening visit and a 4-day confinement period. A final follow up end-of-study telephone call will be performed within a week of last product use.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 18.0 and ≤ 30.0 kg/m2
* Clinically normal medical history
* User of snus or nicotine pouches for ≥1 year, with a minimum weekly use of 2 or more snus or nicotine pouch cans and who is willing and considered able to use brands with nicotine content in the range of 14 to 20 mg nicotine/pouch

Exclusion Criteria:

* History of any clinically significant disease or disorder
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first use of IP.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and HIV
* Female subjects who are pregnant or breastfeeding
* Presence or history of drug or alcohol abuse
* Excessive caffeine consumption defined by a daily intake of >5 cups of caffeine containing beverages
* Intend to change nicotine-use habit or make a quit attempt within the next 3 months from the screening visit.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden

REFERENCES:
- [Derived] Chapman F, Morrissey R, McDermott S, Cahours X, Verron T, Taverner V, Stevenson M, Nahde T. Evaluation of high-nicotine oral products shows potential to reduce tobacco-related harm by offering satisfying alternatives. Sci Rep. 2025 Oct 3;15(1):34636. doi: 10.1038/s41598-025-21812-x. PMID 41044396

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Product Sequence ABCD | Product Sequence BCDA | Product Sequence CDAB | Product Sequence DABC
Started | 7 | 7 | 7 | 6
Completed | 7 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Product Sequence ABCD | Product Sequence BCDA | Product Sequence CDAB | Product Sequence DABC | Total
Number analyzed (Participants) | 7 | 7 | 7 | 6 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (10.2) | 32.4 (14.4) | 30.1 (10.0) | 32.5 (15.0) | 31.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 4 | 2 | 11
  Male | 3 | 6 | 3 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 7 | 6 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 6 | 5 | 5 | 6 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Nicotine Cmax
Description: Maximum observed plasma nicotine concentration
Time Frame: 5 minutes prior to product use and 5, 10, 15, 20, 25, 30, 45, 60, 90 minutes, 2, 4, 6 and 8 hours post start of product use
Population: The analysis population represents all subjects who used a specific product. The overall number of participants analyzed for each product is therefore different from the number of participants in each arm provided in the Participant Flow module.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Product A: All subjects further to use of Product A
- Product B: All subjects further to use of Product B
- Product C: All subjects further to use of Product C
- Product D: All subjects further to use of Product D
Arm/Group | Product A | Product B | Product C | Product D
Number analyzed (Participants) | 27 | 26 | 26 | 27
ng/mL | 14.98 (4.96) | 13.43 (4.97) | 19.35 (6.58) | 13.85 (3.85)

2. Primary Outcome: Nicotine AUCt
Description: The area under the concentration-time curve for nicotine, from time 0 to the time of the last sampling timepoint
Time Frame: 5 minutes prior to product use and at 5, 10, 15, 20, 25, 30, 45, 60, 90 minutes, 2, 4, 6 and 8 hours post start of product use
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Product A | Product B | Product C | Product D
Number analyzed (Participants) | 27 | 26 | 26 | 27
h*ng/mL | 36.48 (12.72) | 31.72 (9.50) | 48.44 (19.68) | 32.11 (9.46)

3. Secondary Outcome: Orally Extracted Amount of Nicotine
Description: Orally extracted fraction of nicotine (%) in the pouch after the 20-minute use period.
Time Frame: 20 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of nicotine
Arm/Group | Product A | Product B | Product C | Product D
Number analyzed (Participants) | 27 | 27 | 27 | 27
Percentage of nicotine | 19.10 (9.98) | 22.9 (10.3) | 21.9 (9.77) | 14.0 (4.63)

4. Secondary Outcome: Urge to Use Emax
Description: The subjects will self-assess their urge to use a nicotine pouch, pre-use and after use, by answering the question: "How strong is your urge to use a nicotine pouch right now?" on a 100 mm visual analogue scale (VAS), with the anchor points 0 mm (= not at all/no urge) and 100 mm (= extremely/extreme urge). Emax is the maximum change from baseline VAS score (VASpre-use - VASpost-use).
Time Frame: 5 minutes prior to product use and at 5, 10, 15, 20, 25, 30, 45 minutes, and 1, 1.5, 2, 4, 6 and 8 hours post start of product use
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Product A | Product B | Product C | Product D
Number analyzed (Participants) | 27 | 27 | 25 | 26
mm | 61.7 (23.3) | 57.7 (19.7) | 66.1 (22.4) | 52.7 (25.7)

ADVERSE EVENTS:
Time Frame: 7 days
Description: The number of participants at risk represents all subjects who used a specific product. The overall number of participants analyzed for each product is therefore different from the number of participants in each arm provided in the Participant Flow module.
Arm/Group | Product A | Product B | Product C | Product D
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 2/27 | 6/27 | 1/27 | 3/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Product A (N=27) | Product B (N=27) | Product C (N=27) | Product D (N=27)
Photophobia (Eye disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 4 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT05452278/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT05452278/SAP_001.pdf